CLINICAL TRIAL: NCT05293509
Title: Pharmacologic Pretransplant Immunosuppression (PTIS) + Reduced Toxicity Conditioning (RTC) Allogeneic Stem Cell Transplantation in Inherited Hematologic Disorders
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0477; NCI-2022-02150 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Stem Cell Transplantation
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Dexamethasone; Cyclophosphamide; Bortezomib; Rituximab; Busulfan; Tacrolimus; Cyclosporine; Mycophenolic Acid; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I: Sequential Pharmacological PTIS (Experimental)
  Interventions: Drug: Fludarabine; Drug: Dexamethasone; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Rituximab; Drug: Busulfan; Drug: Cyclophosphamide (Cy); Drug: Tacrolimus (or cyclosporine)
- Phase II: RTC Regimen and GVHD Prophylaxis Based on Post-Cy (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Busulfan; Drug: Cyclophosphamide (Cy); Drug: Tacrolimus (or cyclosporine); Drug: Mycophenolate mofetil (MMF); Drug: Rabbit ATG

INTERVENTIONS:
Drug: Fludarabine — 40 mg/m2/day i.v.- by vein
  Other Names: Fludara™
Drug: Dexamethasone — 25 mg/m2/day i.v.-by vein
  Arms: Phase I: Sequential Pharmacological PTIS
Drug: Cyclophosphamide — 100 mg/m2 IV-by vein
  Other Names: Cytoxan™
Drug: Bortezomib — Four doses of bortezomib at a dose of 1.3 mg/m2 -injection under the skin
  Other Names: Velcade®
  Arms: Phase I: Sequential Pharmacological PTIS
Drug: Rituximab — Four doses of rituximab at a dose of 375 mg/m2- by vein
  Other Names: Rituxan®
  Arms: Phase I: Sequential Pharmacological PTIS
Drug: Busulfan — 110 mg/m2 i.v-by vein
  Other Names: Busulfex™
Drug: Cyclophosphamide (Cy) — by vein
  Other Names: Cytoxan™
Drug: Tacrolimus (or cyclosporine) — by vein
Drug: Mycophenolate mofetil (MMF) — given by PO
  Arms: Phase II: RTC Regimen and GVHD Prophylaxis Based on Post-Cy
Drug: Rabbit ATG — by vein
  Arms: Phase II: RTC Regimen and GVHD Prophylaxis Based on Post-Cy

SUMMARY:
To assess the outcomes of NRM when administering pharmacologic pretransplant immunosuppression (PTIS) followed by pretransplant reduced toxicity conditioning (RTC) and an allogeneic stem cell transplant (allo-SCT) and post-transplant graft-versus-host disease prophylaxis based on post-transplant cyclophosphamide (PT-Cy) in patients with inherited blood disorders.

DETAILED DESCRIPTION:
Objectives

Primary:

To estimate the 100-day non-relapse mortality (NRM) rate when administering pharmacologic pretransplant immunosuppression (PTIS) followed by pretransplant reduced toxicity conditioning (RTC) and an allogeneic stem cell transplant (allo-SCT) and post-transplant graft-versus-host disease prophylaxis based on post-transplant cyclophosphamide (PT-Cy) in patients with inherited blood disorders.

Secondary outcomes include the following:

i. Immune reconstitution ii. Infectious complications iii. Quality of life (QOL) at 3 months,100 days, and 1 year post-transplant iv. OS, EFS, and GRFS v. Incidence of aGVHD at day 100. vi. Rate of chronic GVHD within the first-year post transplantation. vii. Rate of Graft failure

ELIGIBILITY:
Inclusion Criteria:

1. The first six patients will be ages >12 years old and <35 years old. Thereafter in a second stage, patients ages 2 to 50 years old will be included.
2. Patient with a matched related donor or who has a related haploidentical donor identified.
3. Performance score of at least 70 by Karnofsky or 0 to 1 by ECOG (age > 12 years), or Zubrod or Lansky Play Performance Scale of at least 70 (age <12 years).
4. Adequate major organ system function as demonstrated by:

   1. Serum creatinine clearance equal or more than 50 ml/min (calculated with Cockroft-Gault formula).
   2. Bilirubin equal or less than 1.5 mg/dl except for Gilbert's disease. ALT and/or AST equal or less than 3x institutional ULN. Conjugated (direct) bilirubin less than 2x upper limit of normal.
   3. Left ventricular ejection fraction equal or greater than 50%.
   4. Diffusing capacity for carbon monoxide (DLCO) equal or greater than 50%
   5. Predicted, corrected for hemoglobin. For children < 7 years of age who are unable to perform PFT, oxygen saturation > 92% on room air by pulse oximetry.
5. Patient or the patient's legal representative, parent(s) or guardian should be able to provide written informed consent. Assent of a minor if participant's age is at least seven and less than eighteen years.
6. Sexually active males and females of childbearing potential must agree to use a form of contraception considered effective and medically acceptable by the Investigator.

Exclusion Criteria:

1. HIV positive; active hepatitis B or C.
2. Uncontrolled infections.
3. Liver cirrhosis. However mild fibrosis will be allowed i.e. fine reticulin or Grade 1, with bridging fibrosis.
4. CNS involvement within 3 months.
5. Positive pregnancy test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
6. Inability to comply with medical therapy or follow-up.
7. Will restrict eligibility to a maximum BMI of ≤40
8. Patient with a known history of allergic reactions to any constituents of the cell product, including a known history of allergic reactions to DMSO.
9. Prior allo-SCT
10. Other active malignancy/cancer diagnosis in remission for at least 2yrs. Malignancies not being excluded are as follows: Ductal carcinoma in situ (DCIS), Basal cell carcinoma (BCC), Cervical intraepithelial neoplasia (CIN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
To determine the 100-day non-relapse mortality (NRM) rate when administering pharmacologic pretransplant immunosuppression (PTIS) followed by pretransplant reduced toxicity conditioning (RTC | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Ramdial, Ramdial, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org